CLINICAL TRIAL: NCT02253173
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multi-center Trial to Evaluate the Safety and Efficacy of TX-004HR in Postmenopausal Women With Moderate to Severe Symptoms of Vulvar and Vaginal Atrophy
Brief Title: Estradiol Vaginal Softgel Capsules in Treating Symptoms of Vulvar and Vaginal Atrophy in Postmenopausal Women
Acronym: REJOICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXV14-01
Record Dates: First submitted 2014-09-26; First posted 2014-10-01 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Vulvovaginal Atrophy; Menopause; Dyspareunia; Painful Intercourse
Keywords: VVA; Painful Sex; Postmenopausal
MeSH Terms: conditions — Dyspareunia | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Estradiol 4mcg Vaginal Softgel Capsule (Experimental): Estradiol 4mcg Vaginal Softgel Capsule
  Interventions: Drug: Estradiol
- Estradiol 10mcg Vaginal Softgel Capsule (Experimental): Estradiol 10mcg Vaginal Softgel Capsule
  Interventions: Drug: Estradiol
- Estradiol 25mcg Vaginal Softgel Capsule (Experimental): Estradiol 25mcg Vaginal Softgel Capsule
  Interventions: Drug: Estradiol
- Placebo Vaginal Softgel Capsule (Placebo Comparator): Placebo Vaginal Softgel Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol
  Arms: Estradiol 10mcg Vaginal Softgel Capsule; Estradiol 25mcg Vaginal Softgel Capsule; Estradiol 4mcg Vaginal Softgel Capsule
Drug: Placebo
  Arms: Placebo Vaginal Softgel Capsule

SUMMARY:
This study will assess the safety and efficacy of a new formulation of vaginal estradiol for the treatment of symptoms of vulvar and vaginal atrophy in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female subjects between the ages of 40 and 75 years (at the time of randomization) with at least:

   * 12 months of spontaneous amenorrhea (women <55 years of age with a history of hysterectomy without bilateral oophorectomy prior to natural menopause must have follicle stimulating hormone (FSH) levels > 40 mIU/mL), OR
   * 6 months of spontaneous amenorrhea with follicle stimulating hormone (FSH) levels > 40mlU/mL OR
   * At least 6 weeks postsurgical bilateral oophorectomy.
2. ≤5% superficial cells on vaginal cytological smear
3. Vaginal pH > 5.0
4. Moderate to severe symptom of vaginal pain associated with sexual activity considered the most bothersome vaginal symptom by the subject at screening visit 1A.
5. Moderate to severe symptom of vaginal pain associated with sexual activity at screening visit 1B.
6. Onset of moderate to severe dyspareunia in the postmenopausal years.
7. Subjects should be sexually active (i.e. have sexual activity with vaginal penetration within approximately 1 month of screening visit 1A).
8. Subjects should anticipate having sexual activity (with vaginal penetration) during the conduct of the trial.
9. For subjects with an intact uterus: Subjects must have an acceptable result from an evaluable screening endometrial biopsy.
10. Subjects who have a Body Mass Index (BMI) less than or equal to 38 kg/m2. BMI values should be rounded to the nearest integer (ex. 32.4 rounds down to 32, while 26.5 rounds up to 27).
11. In the opinion of the investigator, the subject will comply with the protocol and has a high probability of completing the study.

Exclusion Criteria:

1. Use of the following:

   1. Oral estrogen-, progestin-, androgen-, or SERM-containing drug products within 8 weeks before screening visit 1A (can enter washout);
   2. Use of transdermal hormone products within 4 weeks before screening visit 1A (can enter washout);
   3. Use of vaginal hormone products (rings, creams, gels) within 4 weeks before screening visit1A (can enter washout);
   4. Use of intrauterine progestins within 8 weeks before screening visit 1A (can enter washout);
   5. Use of progestin implants/injectables or estrogen pellets/injectables within 6 months before screening visit 1A (cannot enter washout);
   6. Use of vaginal lubricants or moisturizers within 7 days before the screening visit 1B vaginal pH assessment.
2. A history or active presence of clinically important medical disease that might confound the study or be detrimental to the subject, examples include:

   1. Hypersensitivity to estrogens;
   2. Endometrial hyperplasia;
   3. Undiagnosed vaginal bleeding;
   4. Have a history of a chronic liver or kidney dysfunction/disorder (e.g., Hepatitis C or chronic renal failure);
   5. Thrombophlebitis, thrombosis or thromboembolic disorders;
   6. Cerebrovascular accident, stroke, or transient ischemic attack;
   7. Myocardial infarction or ischemic heart disease;
   8. Malignancy or treatment for malignancy, within the previous 5 years, with the exception of basal cell carcinoma of the skin or squamous cell carcinoma of the skin. A history of estrogen dependent neoplasia, breast cancer, melanoma or any gynecologic cancer, at any time, excludes the subject;
   9. Endocrine disease (except for controlled hypothyroidism or controlled non-insulin dependent diabetes mellitus).
3. Recent history of known alcohol or drug abuse.
4. History of sexual abuse or spousal abuse that, in the opinion of the PI, may interfere with the subject's assessment of vaginal pain with sexual activity.
5. Current history of Heavy smoking (more than 15 cigarettes per day) or use of e-cigarettes.
6. Use of an intrauterine device within 12 weeks before screening visit 1A.
7. Use of an investigational drug within 60 days before screening visit 1A.
8. Any clinically important abnormalities on screening physical exam, assessments, ECG, or laboratory tests, such as:

   1. Unresolved cervical cytologic smear report of atypical glandular cells of undetermined significance (AGUS) or atypical squamous cells of undetermined significance (ASCUS).

      Cervical cytologic smear report of low-grade squamous intraepithelial lesion (SIL) or greater, CIN1 or greater, or any reported dysplasia; Subjects with ASCUS are eligible only if high risk human papilloma virus (HPV) result is negative.
   2. Unresolved findings suspicious for malignancy on the breast exam; incomplete mammogram result (BI-RADS 0) or unresolved findings suggestive of malignant changes or findings requiring short interval follow-up on the prestudy mammogram (subjects must have mammography result of BI-RADS 1 or 2 to enroll.) Mammogram may be performed within 9 months prior to Visit 2 (randomization) with documentation available. (The site must obtain a copy of the official report for the subject's study file, and it must be verified that the mammogram itself is available if needed for additional assessment);
   3. In subjects with intact uterus: have a screening endometrial biopsy sample that is found by both primary pathologists to have endometrial tissue insufficient for diagnosis, no endometrium identified, or no tissue identified. (With the approval of the Medical Monitor, the screening endometrial biopsy may be repeated once);
   4. In subjects with intact uterus: an endometrial biopsy report by one central pathologist at screening with one of the following:

      * Endometrial hyperplasia endometrial cancer, proliferative endometrium, weakly proliferative endometrium, disordered proliferative pattern; OR
      * Endometrial polyps with hyperplasia, glandular atypia of any degree (e.g., atypical nuclei) or cancer;
   5. Vulvar or vaginal inflammatory condition such as a contact or allergic dermatitis, lichen sclerosis or other pathological findings;
   6. Presence of suspicious vulvar or vaginal lesions for dysplasia, malignancy or other pathology other than atrophy;
   7. Painful genital warts or localized areas of ulceration;
   8. A history of active, chronic pelvic pain;
   9. Interstitial cystitis;
   10. Serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) greater than 1.5 times the upper limit of normal for the laboratory used;
   11. Fasting total cholesterol greater than 300 mg/dL (7.77 mmol/L) or triglycerides greater than 300 mg/dL (3.39 mmol/L);
   12. Fasting blood glucose greater than 125 mg/dL (6.94 mmol/L) with a hemoglobin A1C of greater than or equal to 6.5%;
   13. Uncontrolled hypertension; subjects with elevated sitting blood pressure, greater than 140 mm Hg systolic or greater than 90 mm Hg diastolic and may not be using more than 2 antihypertensive medications for the treatment of hypertension;
   14. Clinically significant abnormal 12-lead ECG (such as myocardial infarction or other findings suggestive of ischemia)
9. Be known to be pregnant or have a positive urine pregnancy test. (Note: A pregnancy test is not required for subjects who have had bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or are 55 years old or greater and have experienced cessation of menses for at least 1 year.
10. Current use of marijuana.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (105):
- United States (100):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Montogomery Women's Health, Montgomery, Alabama
  - Cactus Clinical Research, Mesa, Arizona
  - Arizona Wellness Center for Women, Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Sutter East Bay Medical Foundation, Berkeley, California
  - Torrance Clinical Research Institute Inc, Lomita, California
  - Futura Research, Norwalk, California
  - Northern California Research, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - San Diego Sexual Medicine, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clinical Research Center, Denver, Colorado
  - Red Rocks OB/Gyn, Lakewood, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - James A. Simon, Women's Health & Research Consultants, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Avail Clinical Research, DeLand, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - UF Health Physicians Women's & REI Springhill, Gainesville, Florida
  - UF College of Medicine-Jacksonville, Dept. of Obstetrics and Gynecology, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - South Florida Wellness & Clinical Research Institute, Margate, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Healthcare Clinical Data, North Miami, Florida
  - Ideal Clinical Research, North Miami Beach, Florida
  - Radiant Research, Pinellas Park, Florida
  - All Women's Healthcare of West Broward, Plantation, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Women's Health Associates, Atlanta, Georgia
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - WR-Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Women's Healthcare Associates P.A., Idaho Falls, Idaho
  - Radiant Research, Chicago, Illinois
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Lafayette Clinical Research Group, Lafayette, Indiana
  - Cypress Medical Research Center, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Horizon Research Group of Opelousas, Eunice, Louisiana
  - Capital Women's Care, Frederick, Maryland
  - Maryland Center for Sexual Health, Lutherville, Maryland
  - ClinSite, LLC, Ann Arbor, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Saginaw Valley Medical Research Group, L.L.C., Saginaw, Michigan
  - Montana Health, Billings, Montana
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Office of Edmond E. Pack, MD, Las Vegas, Nevada
  - Office of R. Garn Mabey, MD, Las Vegas, Nevada
  - Lawrence OB-GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Bosque Women's Care, Albuquerque, New Mexico
  - Southwest Clinical Research, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Suffolk OB/GYN, Port Jefferson, New York
  - Women's Wellness Clinic, Durham, North Carolina
  - Pinewest OB-GYN, Inc., High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hawthorne Research, Winston-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Radiant Research, Akron, Ohio
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Landerbrook Health Center, Mayfield Heights, Ohio
  - Sunstone Medical Research, Medford, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - Vista Clinical Research, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Research Across America, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Advances in Health, Houston, Texas
  - Hwca, Pllc, Houston, Texas
  - TMC Life Research, Houston, Texas
  - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - National Clinical Research-Norfolk, Norfolk, Virginia
  - Clinical Research Center, EVMS, Norfolk, Virginia
  - Virginia Women's Center, Inc., Richmond, Virginia
  - National Clinical Research-Richmond, Inc, Richmond, Virginia
  - Tidewater Clinical Research, Virginia Beach, Virginia
  - Seattle Women's Health, Research, and Gynecology, Seattle, Washington
  - North Spokane Women's Health, Spokane, Washington
- Canada (5):
  - Diex Research Montreal Inc., Montreal, Quebec
  - Center for Research Saint-Louis, Québec, Quebec
  - Manna Research Inc, Saint Romuald, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Clinique RSF Inc., Québec

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252
- [Derived] Mirkin S, Simon JA, Liu JH, Archer DF, Castro PD, Graham S, Bernick B, Komm B. Evaluation of endometrial progesterone receptor expression after 12 weeks of exposure to a low-dose vaginal estradiol insert. Menopause. 2021 May 28;28(9):998-1003. doi: 10.1097/GME.0000000000001801. PMID 34054104
- [Derived] Constantine G, Millheiser LS, Kaunitz AM, Parish SJ, Graham S, Bernick B, Mirkin S. Early onset of action with a 17beta-estradiol, softgel, vaginal insert for treating vulvar and vaginal atrophy and moderate to severe dyspareunia. Menopause. 2019 Nov;26(11):1259-1264. doi: 10.1097/GME.0000000000001394. PMID 31688572
- [Derived] Constantine GD, Simon JA, Pickar JH, Archer DF, Bernick B, Graham S, Mirkin S. Estradiol vaginal inserts (4 microg and 10 microg) for treating moderate to severe vulvar and vaginal atrophy: a review of phase 3 safety, efficacy and pharmacokinetic data. Curr Med Res Opin. 2018 Dec;34(12):2131-2136. doi: 10.1080/03007995.2018.1527578. Epub 2018 Sep 28. PMID 30238814
- [Derived] Constantine GD, Bouchard C, Pickar JH, Archer DF, Graham S, Bernick B, Mirkin S. Consistency of Effect with a Low-Dose, Estradiol Vaginal Capsule (TX-004HR): Evaluating Improvement in Vaginal Physiology and Moderate-to-Severe Dyspareunia in Subgroups of Postmenopausal Women. J Womens Health (Larchmt). 2017 Jun;26(6):616-623. doi: 10.1089/jwh.2016.6187. Epub 2017 Mar 29. PMID 28355090

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol 4mcg Vaginal Softgel Capsule: Estradiol 4mcg Vaginal Softgel Capsule
  Estradiol
- Estradiol 10mcg Vaginal Softgel Capsule: Estradiol 10mcg Vaginal Softgel Capsule
  Estradiol
- Estradiol 25mcg Vaginal Softgel Capsule: Estradiol 25mcg Vaginal Softgel Capsule
  Estradiol
- Placebo Vaginal Softgel Capsule: Placebo Vaginal Softgel Capsule
  Placebo
Period: Overall Study
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Started | 191 | 191 | 190 | 192
Completed | 175 | 174 | 177 | 178
Not Completed | 16 | 17 | 13 | 14

BASELINE CHARACTERISTICS:
Population: The modified intent to treat (MITT) population was the primary efficacy population, defined as all ITT subjects who received the treatment to which they were randomized, had baseline values for all co-primary variables, and had at least one post-baseline value for any of the four co-primary variables at any visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule | Total
Number analyzed (Participants) | 191 | 191 | 190 | 192 | 764
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 148 | 162 | 156 | 151 | 617
  >=65 years | 43 | 29 | 34 | 41 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (5.90) | 58.5 (6.29) | 58.9 (6.26) | 59.3 (6.07) | 59.1 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 191 | 190 | 192 | 764
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 10 | 15 | 12 | 50
  United States | 178 | 181 | 175 | 180 | 714
Height [Mean (Standard Deviation); unit: centimeters] | 162.7 (6.86) | 162.9 (6.93) | 162.3 (6.37) | 162.2 (6.30) | 162.5 (6.62)
Weight [Mean (Standard Deviation); unit: kilograms] | 70.4 (14.26) | 71.1 (13.49) | 70.6 (13.7) | 70.4 (13.6) | 70.6 (13.74)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.87) | 26.8 (4.68) | 26.7 (4.79) | 26.7 (4.59) | 26.7 (4.73)

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Efficacy Endpoint - Vaginal Superficial Cells
Description: • Change from Baseline to Week 12 in the percentage of vaginal superficial cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and 12 Weeks
Population: For the statistical test utilized (MMRM), the number of subjects analyzed varied based on if they had both Baseline and Week 12 data so it would not necessarily match the overall number of subjects in the MITT Population at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal superficial cells
Groups:
- Estradiol 4mcg Vaginal Softgel Capsule; Estradiol 10mcg Vaginal Softgel Capsule; Estradiol 25mcg Vaginal Softgel Capsule; Placebo: Postmenopausal women self-administered intravaginally one capsule daily for 14 days and then bi-weekly for 10 weeks.
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo
Number analyzed (Participants) | 170 | 171 | 174 | 172
percentage of vaginal superficial cells | 17.50 (1.542) | 16.72 (1.540) | 23.20 (1.529) | 5.63 (1.537)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

2. Primary Outcome: Co-Primary Efficacy Endpoint - Vaginal Parabasal Cells
Description: • Change from Baseline to Week 12 in the percentage of vaginal parabasal cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal parabasal cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo
Number analyzed (Participants) | 170 | 171 | 174 | 172
percentage of vaginal parabasal cells | -40.63 (1.755) | -44.07 (1.751) | -45.55 (1.745) | -6.73 (1.750)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

3. Primary Outcome: Co-Primary Efficacy Endpoint - Vaginal pH
Description: • Change from Baseline to Week 12 in vaginal pH as compared to placebo
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pH units
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo
Number analyzed (Participants) | 170 | 171 | 174 | 174
pH units | -1.32 (0.066) | -1.42 (0.066) | -1.34 (0.066) | -0.28 (0.066)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

4. Primary Outcome: Co-Primary Efficacy Endpoint - Severity of Most Bothersome Symptom (Dyspareunia)
Description: • Change from Baseline to Week 12 on the severity of the MBS of dyspareunia (vaginal pain associated with sexual activity) associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo
Number analyzed (Participants) | 151 | 154 | 159 | 163
units on a scale | -1.52 (0.071) | -1.69 (0.071) | -1.69 (0.071) | -1.28 (0.070)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

5. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Superficial Cells
Description: • Change from Baseline to Week 2 in the percentage of vaginal superficial cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 2
Population: For the statistical test utilized (MMRM), the number of subjects analyzed varied based on if they had both Baseline and Week 2 data so it would not necessarily match the overall number of subjects in the MITT Population at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal superficial cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 186 | 188 | 184 | 185
percentage of vaginal superficial cells | 31.35 (1.496) | 31.93 (1.488) | 38.85 (1.500) | 6.05 (1.498)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

6. Secondary Outcome: Secondary Efficacy Endpoints- Vaginal Superficial Cells
Description: Change from Baseline to Week 6 in the percentage of vaginal superficial cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 6
Population: For the statistical test utilized (MMRM), the number of subjects analyzed varied based on if they had both Baseline and Week 6 data so it would not necessarily match the overall number of subjects in the MITT Population at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal superficial cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
percentage of vaginal superficial cells | 18.41 (1.536) | 16.88 (1.543) | 22.65 (1.532) | 5.43 (1.525)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

7. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Superficial Cells
Description: Change from Baseline to Week 8 in the percentage of vaginal superficial cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 8
Population: For the statistical test utilized (MMRM), the number of subjects analyzed varied based on if they had both Baseline and Week 8 data so it would not necessarily match the overall number of subjects in the MITT Population at Baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal superficial cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
percentage of vaginal superficial cells | 19.04 (1.561) | 17.41 (1.558) | 23.88 (1.554) | 5.98 (1.551)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

8. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Parabasal Cells
Description: Change from Baseline to Week 2 in the percentage of vaginal parabasal cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal parabasal cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 186 | 188 | 184 | 185
percentage of vaginal parabasal cells | -40.23 (1.720) | -44.42 (1.710) | -45.60 (1.723) | -7.00 (1.720)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

9. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Parabasal Cells
Description: Change from Baseline to Week 6 in the percentage of vaginal parabasal cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal parabasal cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
percentage of vaginal parabasal cells | -39.36 (1.750) | -43.55 (1.752) | -45.61 (1.746) | -9.23 (1.741)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

10. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Parabasal Cells
Description: Change from Baseline to Week 8 in the percentage of vaginal parabasal cells (by vaginal cytologic smear) compared to placebo
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percentage of vaginal parabasal cells
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
percentage of vaginal parabasal cells | -41.87 (1.768) | -43.78 (1.764) | -45.08 (1.762) | -7.86 (1.760)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

11. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal pH
Description: Change from Baseline to Week 2 in vaginal pH as compared to placebo
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: pH units
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 186 | 188 | 184 | 186
pH units | -1.23 (0.064) | -1.37 (0.064) | -1.30 (0.065) | -0.28 (0.064)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

12. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal pH
Description: Change from Baseline to Week 6 in vaginal pH as compared to placebo
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: pH units
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
pH units | -1.32 (0.066) | -1.40 (0.066) | -1.48 (0.066) | -0.30 (0.065)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

13. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal pH
Description: Change from Baseline to Week 8 in vaginal pH as compared to placebo
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: pH units
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
pH units | -1.35 (0.067) | -1.46 (0.067) | -1.45 (0.066) | -0.38 (0.066)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

14. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Most Bothersome Symptom (Dyspareunia)
Description: Change from Baseline to Week 2 on the severity of the MBS of dyspareunia (vaginal pain associated with sexual activity) associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 145 | 147 | 140 | 141
units on a scale | -0.99 (0.072) | -1.08 (0.072) | -1.02 (0.073) | -0.76 (0.072)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0260, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0105, Mixed Models Analysis

15. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Most Bothersome Symptom (Dyspareunia)
Description: Change from Baseline to Week 6 on the severity of the MBS of dyspareunia (vaginal pain associated with sexual activity) associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 148 | 150 | 150 | 159
units on a scale | -1.30 (0.072) | -1.37 (0.072) | -1.48 (0.072) | -1.03 (0.070)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

16. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Most Bothersome Symptom (Dyspareunia)
Description: Change from Baseline to Week 8 on the severity of the MBS of dyspareunia (vaginal pain associated with sexual activity) associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 140 | 136 | 129 | 143
units on a scale | -1.52 (0.073) | -1.64 (0.074) | -1.62 (0.075) | -1.15 (0.072)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

17. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Other VVA Symptoms (Vaginal Dryness)
Description: Change from Baseline to Week 2 on the severity of vaginal dryness associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 186 | 188 | 184 | 185
units on a scale | -0.86 (0.066) | -1.01 (0.065) | -0.96 (0.066) | -0.72 (0.066)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.1269, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0082, Mixed Models Analysis

18. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Other VVA Symptoms (Vaginal Dryness)
Description: Change from Baseline to Week 6 on the severity of vaginal dryness associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 172 | 176
units on a scale | -1.14 (0.067) | -1.27 (0.068) | -1.23 (0.067) | -0.90 (0.067)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis

19. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Other VVA Symptoms (Vaginal Dryness)
Description: Change from Baseline to Week 8 on the severity of vaginal dryness associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 163 | 165 | 165 | 167
units on a scale | -1.25 (0.069) | -1.44 (0.068) | -1.34 (0.068) | -1.01 (0.068)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis

20. Secondary Outcome: Secondary Efficacy Endpoints - Severity of Other VVA Symptoms (Vaginal Dryness)
Description: Change from Baseline to Week 12 on the severity of vaginal dryness associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 176 | 174
units on a scale | -1.27 (0.068) | -1.47 (0.067) | -1.47 (0.067) | -0.97 (0.067)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

21. Secondary Outcome: Secondary Efficacy Endpoints - Other VVA Symptoms (Vulvar and/or Vaginal Itching or Irritation)
Description: Change from Baseline to Week 2 on the severity of vulvar and/or vaginal itching or irritation associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 186 | 188 | 184 | 185
units on a scale | -0.47 (0.054) | -0.56 (0.053) | -0.51 (0.054) | -0.47 (0.054)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9616, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.2439, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.6518, Mixed Models Analysis

22. Secondary Outcome: Secondary Efficacy Endpoints - Other VVA Symptoms (Vulvar and/or Vaginal Itching or Irritation)
Description: Change from Baseline to Week 6 on the severity of vulvar and/or vaginal itching or irritation associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 172 | 176
units on a scale | -0.57 (0.055) | -0.64 (0.055) | -0.61 (0.055) | -0.55 (0.055)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.7829, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.2328, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.4118, Mixed Models Analysis

23. Secondary Outcome: Secondary Efficacy Endpoints - Other VVA Symptoms (Vulvar and/or Vaginal Itching or Irritation)
Description: Change from Baseline to Week 8 on the severity of vulvar and/or vaginal itching or irritation associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 163 | 165 | 165 | 167
units on a scale | -0.74 (0.056) | -0.76 (0.056) | -0.73 (0.056) | -0.59 (0.056)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0639, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0356, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0914, Mixed Models Analysis

24. Secondary Outcome: Secondary Efficacy Endpoints - Other VVA Symptoms (Vulvar and/or Vaginal Itching or Irritation)
Description: Change from Baseline to Week 12 on the severity of vulvar and/or vaginal itching or irritation associated with VVA as compared to placebo
  VVA Symptoms Self-Assessment Questionnaire Severity Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe.
  Subjects assessed severity at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 176 | 174
units on a scale | -0.75 (0.055) | -0.81 (0.055) | -0.77 (0.055) | -0.60 (0.055)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0503, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0263, Mixed Models Analysis

25. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Color)
Description: Change from Baseline to Week 2 in Vaginal Color as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Color: No atrophy (pink) = 0; Mild (lighter in color) = 1; Moderate(pale in color) = 2; Severe (transparent/no color or inflamed) = 3 Severity was assessed by the Investigator at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 185 | 187 | 184 | 187
units on a scale | -0.69 (0.048) | -0.77 (0.047) | -0.78 (0.048) | -0.40 (0.047)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

26. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Color)
Description: Change from Baseline to Week 6 in Vaginal Color as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Color: No atrophy (pink) = 0; Mild (lighter in color) = 1; Moderate(pale in color) = 2; Severe (transparent/no color or inflamed) = 3 Severity was assessed by the Investigator at Baseline and Week 6
Time Frame: Baseline to Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
units on a scale | -0.82 (0.049) | -0.93 (0.049) | -0.89 (0.049) | -0.50 (0.048)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

27. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Color)
Description: Change from Baseline to Week 8 in Vaginal Color as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Color: No atrophy (pink) = 0; Mild (lighter in color) = 1; Moderate(pale in color) = 2; Severe (transparent/no color or inflamed) = 3 Severity was assessed by the Investigator at Baseline and Week 8
Time Frame: Baseline to Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
units on a scale | -0.98 (0.050) | -1.04 (0.050) | -0.99 (0.049) | -0.50 (0.049)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

28. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Color)
Description: Change from Baseline to Week 12 in Vaginal Color as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Color: No atrophy (pink) = 0; Mild (lighter in color) = 1; Moderate(pale in color) = 2; Severe (transparent/no color or inflamed) = 3 Severity was assessed by the Investigator at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 175 | 175
units on a scale | -0.97 (0.049) | -1.06 (0.049) | -0.96 (0.049) | -0.60 (0.049)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

29. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Integrity)
Description: Change from Baseline to Week 2 in Vaginal Epithelial Integrity as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Integrity: No atrophy (normal) = 0; Mild (vaginal surface bleeds with scraping) = 1; Moderate (vaginal surface bleeds with light contact) = 2; Severe (vaginal surface has petechiae before contact and bleeds with light contact) = 3
  Severity was assessed by the Investigator at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 185 | 187 | 184 | 186
units on a scale | -0.85 (0.049) | -0.87 (0.049) | -0.93 (0.049) | -0.53 (0.049)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

30. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Integrity)
Description: Change from Baseline to Week 6 in Vaginal Epithelial Integrity as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Integrity: No atrophy (normal) = 0; Mild (vaginal surface bleeds with scraping) = 1; Moderate (vaginal surface bleeds with light contact) = 2; Severe (vaginal surface has petechiae before contact and bleeds with light contact) = 3
  Severity was assessed by the Investigator at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
units on a scale | -0.97 (0.051) | -1.02 (0.051) | -1.01 (0.051) | -0.61 (0.050)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

31. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Integrity)
Description: Change from Baseline to Week 8 in Vaginal Epithelial Integrity as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Integrity: No atrophy (normal) = 0; Mild (vaginal surface bleeds with scraping) = 1; Moderate (vaginal surface bleeds with light contact) = 2; Severe (vaginal surface has petechiae before contact and bleeds with light contact) = 3
  Severity was assessed by the Investigator at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
units on a scale | -1.03 (0.052) | -1.08 (0.051) | -1.08 (0.051) | -0.66 (0.051)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

32. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Integrity)
Description: Change from Baseline to Week 12 in Vaginal Epithelial Integrity as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Integrity: No atrophy (normal) = 0; Mild (vaginal surface bleeds with scraping) = 1; Moderate (vaginal surface bleeds with light contact) = 2; Severe (vaginal surface has petechiae before contact and bleeds with light contact) = 3
  Severity was assessed by the Investigator at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 175 | 175
units on a scale | -0.97 (0.051) | -1.07 (0.051) | -1.01 (0.050) | -0.60 (0.050)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

33. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Surface Thickness)
Description: Change from Baseline to Week 2 in Vaginal Epithelial Surface Thickness as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Surface Thickness: No atrophy (rogation and elasticity of vault) = 0; Mild (poor rogation with some elasticity noted of vaginal vault) = 1; Moderate (smooth, some elasticity of vaginal vault) = 2; Severe [smooth, no elasticity, constriction of the upper one third of vagina or loss of vaginal tone (cystocele and rectocele)] = 3
  Severity was assessed by the Investigator at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 185 | 187 | 184 | 186
units on a scale | -0.76 (0.049) | -0.76 (0.049) | -0.76 (0.049) | -0.40 (0.049)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

34. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Surface Thickness)
Description: Change from Baseline to Week 6 in Vaginal Epithelial Surface Thickness as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Surface Thickness: No atrophy (rogation and elasticity of vault) = 0; Mild (poor rogation with some elasticity noted of vaginal vault) = 1; Moderate (smooth, some elasticity of vaginal vault) = 2; Severe [smooth, no elasticity, constriction of the upper one third of vagina or loss of vaginal tone (cystocele and rectocele)] = 3
  Severity was assessed by the Investigator at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
units on a scale | -0.85 (0.051) | -0.93 (0.051) | -0.90 (0.050) | -0.53 (0.050)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

35. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Surface Thickness)
Description: Change from Baseline to Week 8 in Vaginal Epithelial Surface Thickness as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Surface Thickness: No atrophy (rogation and elasticity of vault) = 0; Mild (poor rogation with some elasticity noted of vaginal vault) = 1; Moderate (smooth, some elasticity of vaginal vault) = 2; Severe [smooth, no elasticity, constriction of the upper one third of vagina or loss of vaginal tone (cystocele and rectocele)] = 3
  Severity was assessed by the Investigator at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
units on a scale | -0.96 (0.051) | -1.04 (0.051) | -0.99 (0.051) | -0.59 (0.051)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

36. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Epithelial Surface Thickness)
Description: Change from Baseline to Week 12 in Vaginal Epithelial Surface Thickness as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Epithelial Surface Thickness: No atrophy (rogation and elasticity of vault) = 0; Mild (poor rogation with some elasticity noted of vaginal vault) = 1; Moderate (smooth, some elasticity of vaginal vault) = 2; Severe [smooth, no elasticity, constriction of the upper one third of vagina or loss of vaginal tone (cystocele and rectocele)] = 3
  Severity was assessed by the Investigator at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 175 | 175
units on a scale | -0.98 (0.051) | -1.03 (0.051) | -0.94 (0.050) | -0.61 (0.050)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

37. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Secretions)
Description: Change from Baseline to Week 2 in Vaginal Secretions as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Secretions: No atrophy (normal clear secretions noted on vaginal walls) = 0; Mild (superficial coating of secretions, difficulty with speculum insertion) = 1; Moderate (scant not covering the entire vaginal vault, may need lubrication with speculum insertion to prevent pain) = 2; Severe (none, inflamed, ulceration noted, need lubrication with speculum insertion to prevent pain) = 3
  Severity was assessed by the Investigator at Baseline and Week 2
Time Frame: Baseline and Week 2
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 185 | 187 | 184 | 186
units on a scale | -0.79 (0.050) | -0.83 (0.050) | -0.86 (0.050) | -0.54 (0.050)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

38. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Secretions)
Description: Change from Baseline to Week 6 in Vaginal Secretions as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Secretions: No atrophy (normal clear secretions noted on vaginal walls) = 0; Mild (superficial coating of secretions, difficulty with speculum insertion) = 1; Moderate (scant not covering the entire vaginal vault, may need lubrication with speculum insertion to prevent pain) = 2; Severe (none, inflamed, ulceration noted, need lubrication with speculum insertion to prevent pain] = 3
  Severity was assessed by the Investigator at Baseline and Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 172 | 170 | 173 | 176
units on a scale | -0.90 (0.051) | -0.95 (0.051) | -0.97 (0.051) | -0.60 (0.051)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

39. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Secretions)
Description: Change from Baseline to Week 8 in Vaginal Secretions as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Secretions: No atrophy (normal clear secretions noted on vaginal walls) = 0; Mild (superficial coating of secretions, difficulty with speculum insertion) = 1; Moderate (scant not covering the entire vaginal vault, may need lubrication with speculum insertion to prevent pain) = 2; Severe (none, inflamed, ulceration noted, need lubrication with speculum insertion to prevent pain] = 3
  Severity was assessed by the Investigator at Baseline and Week 8
Time Frame: Baseline and Week 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 164 | 165 | 166 | 167
units on a scale | -1.00 (0.052) | -1.04 (0.052) | -1.06 (0.052) | -0.63 (0.052)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

40. Secondary Outcome: Secondary Efficacy Endpoints - Vaginal Mucosa Assessment (Vaginal Secretions)
Description: Change from Baseline to Week 12 in Vaginal Secretions as compared to placebo
  Vaginal Mucosa Assessment Scale - Vaginal Secretions: No atrophy (normal clear secretions noted on vaginal walls) = 0; Mild (superficial coating of secretions, difficulty with speculum insertion) = 1; Moderate (scant not covering the entire vaginal vault, may need lubrication with speculum insertion to prevent pain) = 2; Severe (none, inflamed, ulceration noted, need lubrication with speculum insertion to prevent pain] = 3
  Severity was assessed by the Investigator at Baseline and Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 171 | 173 | 175 | 175
units on a scale | -1.01 (0.051) | -1.06 (0.051) | -1.04 (0.051) | -0.64 (0.051)
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

41. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) - Total Score
Description: Change from Baseline to Week 12 in FSFI Total Score as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 153 | 152 | 156 | 158
units on a scale | 7.909 [6.748 to 9.070] | 9.431 [8.261 to 10.601] | 10.283 [9.133 to 11.434] | 7.458 [6.315 to 8.602]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9075, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0492, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0019, ANCOVA

42. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Arousal
Description: Change from Baseline to Week 12 in FSFI Domain Score (Arousal) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 154 | 152 | 157 | 159
units on a scale | 0.875 [0.657 to 1.093] | 1.287 [1.066 to 1.507] | 1.392 [1.176 to 1.608] | 0.93 [0.715 to 1.145]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9719, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0614, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0085, ANCOVA

43. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Desire
Description: Change from Baseline to Week 12 in FSFI Domain Score (Desire) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 154 | 152 | 157 | 159
units on a scale | 0.625 [0.471 to 0.779] | 0.800 [0.646 to 0.955] | 0.848 [0.695 to 1.000] | 0.630 [0.479 to 0.782]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9999, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.2855, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.1189, ANCOVA

44. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Lubrication
Description: Change from Baseline to Week 12 in FSFI Domain Score (Lubrication) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 153 | 152 | 156 | 159
units on a scale | 1.834 [1.578 to 2.090] | 2.242 [1.984 to 2.500] | 2.299 [2.045 to 2.553] | 1.595 [1.343 to 1.846]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.4162, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0013, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0003, ANCOVA

45. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Orgasm
Description: Change from Baseline to Week 12 in FSFI Domain Score (Orgasm) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 153 | 152 | 156 | 159
units on a scale | 1.162 [0.903 to 1.421] | 1.274 [1.013 to 1.535] | 1.591 [1.334 to 1.847] | 1.202 [0.948 to 1.457]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9929, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9634, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0898, ANCOVA

46. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Pain
Description: Change from Baseline to Week 12 in FSFI Domain Score (Pain) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 154 | 152 | 156 | 159
units on a scale | 2.173 [1.879 to 2.467] | 2.548 [2.251 to 2.844] | 2.514 [2.222 to 2.805] | 1.930 [1.641 to 2.219]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.5146, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0099, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0150, ANCOVA

47. Secondary Outcome: Secondary Efficacy Endpoints - Female Sexual Function Index (FSFI) Domain Score - Satisfaction
Description: Change from Baseline to Week 12 in FSFI Domain Score (Satisfaction) as compared to placebo
  The FSFI is a brief, multidimensional questionnaire for assessing sexual function in women (Rosen et al., 2000). The questionnaire consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI questionnaire has a minimum total score of 2.0, a maximum score of 36.0 points and was administered at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo Vaginal Softgel Capsule
Number analyzed (Participants) | 154 | 152 | 157 | 158
units on a scale | 1.257 [1.046 to 1.469] | 1.384 [1.170 to 1.597] | 1.629 [1.420 to 1.839] | 1.174 [0.965 to 1.383]
Statistical Analysis 1: Comparison: Estradiol 4mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.9039, ANCOVA
Statistical Analysis 2: Comparison: Estradiol 10mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.3751, ANCOVA
Statistical Analysis 3: Comparison: Estradiol 25mcg Vaginal Softgel Capsule vs Placebo Vaginal Softgel Capsule; Test type: Superiority or Other; p = 0.0073, ANCOVA

48. Other Pre Specified Outcome: PK Substudy - Hormone Concentration Assessments (Serum Estradiol, Estrone and Estrone Conjugates; SHBG)
Description: Blood samples will be obtained from a subset of subjects at pre-selected sites to characterize PK parameters (AUC, tmax, Cmin, Cmax, Cavg) and to measure SHBG
Time Frame: Pre-treatment, Day 2, Weeks 2 and 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Estradiol 4mcg Vaginal Softgel Capsule | Estradiol 10mcg Vaginal Softgel Capsule | Estradiol 25mcg Vaginal Softgel Capsule | Placebo
Serious Adverse Events (participants affected / at risk) | 0/191 | 3/191 | 4/190 | 1/192
Other Adverse Events (participants affected / at risk) | 46/191 | 41/191 | 45/190 | 66/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol 4mcg Vaginal Softgel Capsule (N=191) | Estradiol 10mcg Vaginal Softgel Capsule (N=191) | Estradiol 25mcg Vaginal Softgel Capsule (N=190) | Placebo (N=192)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol 4mcg Vaginal Softgel Capsule (N=191) | Estradiol 10mcg Vaginal Softgel Capsule (N=191) | Estradiol 25mcg Vaginal Softgel Capsule (N=190) | Placebo (N=192)
Nasopharyngitis (Infections and infestations) | 5 | 6 | 7 | 10
Upper respiratory infection (Infections and infestations) | 5 | 6 | 3 | 5
Urinary tract infection (Infections and infestations) | 5 | 5 | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 4 | 8
Headache (Nervous system disorders) | 12 | 14 | 6 | 15
Vaginal discharge (Reproductive system and breast disorders) | 5 | 6 | 4 | 13
Vulvovaginal pruritus (Reproductive system and breast disorders) | 4 | 3 | 7 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other